CLINICAL TRIAL: NCT01567722
Title: Tissue Acquisition for Analysis of Prognostic Factors, Immunology, and Genetic Progression of HIV-1 Associated Malignancies
Brief Title: Collecting and Studying Tissue Samples From Patients With HIV-Associated Malignancies
Status: Terminated | Type: Observational
Why Stopped: Sponsor directive
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); AIDS and Cancer Specimen Resource (Other); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: AMC-083; CDR0000729843 (Other: NCI); U01CA121947 (NIH)
Record Dates: First submitted 2012-03-29; First posted 2012-03-30 (Estimated); Results first posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Lymphoma
Keywords: HIV infection; adult diffuse large cell lymphoma; non-small cell lung cancer; AIDS-related diffuse large cell lymphoma
MeSH Terms: conditions — Lung Neoplasms; Lymphoma; HIV Infections; Lymphoma, Large B-Cell, Diffuse; Carcinoma, Non-Small-Cell Lung | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh-frozen tissue, peripheral blood mononuclear cells, formalin-fixed, paraffin-embedded tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV-positive diffuse large B-cell lymphoma cases: Tissue collection for genomic sequencing from persons with a diagnosis of HIV and diffuse large B-cell lymphoma.
  Interventions: Genetic: DNA analysis; Genetic: RNA analysis; Genetic: gene expression analysis; Genetic: polymorphism analysis; Other: biologic sample preservation procedure; Other: flow cytometry; Other: medical chart review
- HIV-positive lung cancer cases: Tissue collection for genomic sequencing from persons with a diagnosis of HIV and lung cancer.
  Interventions: Genetic: DNA analysis; Genetic: RNA analysis; Genetic: gene expression analysis; Genetic: polymorphism analysis; Other: biologic sample preservation procedure; Other: flow cytometry; Other: medical chart review
- HIV-positive cervical cancer cases: Tissue specimen collection from HIV positive patients with a diagnosis of cervical cancer

INTERVENTIONS:
Genetic: DNA analysis — This sample will be used for germline DNA analysis.
  Groups: HIV-positive diffuse large B-cell lymphoma cases; HIV-positive lung cancer cases
Genetic: RNA analysis — RNA will be sheared, reverse transcribed, and sequenced to assess transcribed sequences.
  Groups: HIV-positive diffuse large B-cell lymphoma cases; HIV-positive lung cancer cases
Genetic: gene expression analysis — Genomic analyses performed on these samples may include, but are not limited to, array-based gene expression profiling, comparative genome hybridization, and single nucleotide polymorphism studies, as well as whole genome sequencing analysis using the most current genomic technology available.
  Groups: HIV-positive diffuse large B-cell lymphoma cases; HIV-positive lung cancer cases
Genetic: polymorphism analysis — Genomic analyses performed on these samples may include, but are not limited to, array-based gene expression profiling, comparative genome hybridization, and single nucleotide polymorphism studies, as well as whole genome sequencing analysis using the most current genomic technology available.
  Groups: HIV-positive diffuse large B-cell lymphoma cases; HIV-positive lung cancer cases
Other: biologic sample preservation procedure — Genomic analyses performed on these samples may include, but are not limited to, array-based gene expression profiling, comparative genome hybridization, and single nucleotide polymorphism studies, as well as whole genome sequencing analysis using the most current genomic technology available.
  Groups: HIV-positive diffuse large B-cell lymphoma cases; HIV-positive lung cancer cases
Other: flow cytometry — Information will include HIV RNA load at time of malignancy diagnosis) and imaging tests, results of the diagnostic tumor biopsy and bone marrow biopsy, and results of flow cytometry, cytogenetics, and molecular studies.
  Groups: HIV-positive diffuse large B-cell lymphoma cases; HIV-positive lung cancer cases
Other: medical chart review — Participants will be followed prospectively to record the types of treatment given, and treatment outcome and toxicity.
  Groups: HIV-positive diffuse large B-cell lymphoma cases; HIV-positive lung cancer cases

SUMMARY:
RATIONALE: Collecting and studying tissue samples from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies collecting tissue samples from patients with HIV-related malignancies.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain high-quality, clinically annotated tissue from patients with human immunodeficiency virus (HIV)-1 malignancy.
* To study clinical, genetic, and immunologic parameters that have prognostic significance and/or are involved in the initiation and progression of HIV-1 malignancies, including complete genomic sequence determination of HIV-associated diffuse large B-cell lymphomas, lung cancer, anal cancer, and cervical cancer.

OUTLINE: This is a multicenter study.

Patients undergo tumor, lymph node, bone marrow, or skin biopsy, and peripheral blood mononuclear cells collection. Samples are submitted to the AIDS Malignancy Consortium (AMC) Biorepository and transferred to the AIDS and Cancer Specimen Resource (ACSR). Samples are then analyzed by the Genome Science Center of British Columbia (GSC-BC) and the HIV+ Tumor Molecular Characterization Project (HTMCP) for full genomic sequencing analysis that may include, but are not limited to, array-based gene expression profiling, comparative genome hybridization, and single nucleotide polymorphism studies by flow cytometry, cytogenetics, and molecular studies. Patients' clinical data, demographics, and treatment given are also collected prospectively in order to record treatment outcome and toxicity.

Patients are followed up at 6 months, 1 year, and 2 years for data-reporting purposes.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Participants must have a diagnosis of a malignancy or clinical findings suggestive of a possible HIV-associated malignancy of one of three types:

  * Diffuse large B-cell lymphoma
  * Non-small cell lung malignancy
* The presence of any of the following conditions will exclude a participant from study enrollment:

  * Absence of sufficient diagnostic tumor-biopsy tissue material to meet the protocol requirements for baseline specimen submission (minimum specimen size of 10 x 10 x 2 mm); repeat tumor biopsy will not be performed solely to meet the protocol specimen-collection requirements
  * Participants whose biopsies, for the purpose of this protocol, show a diagnosis of anal intraepithelial neoplasia or cervical intraepithelial neoplasia
  * Prior treatment for the study malignancy (including neo-adjuvants), since treatment can affect the mutational spectra of tumors
* HIV infection based on serologic documentation of HIV infection at any time prior to study entry, as evidenced by positive enzyme-linked immunosorbent assay (ELISA), positive western blot, or any other Food and Drug Administration (FDA)-approved (licensed) HIV test; alternatively, this documentation may include a record that another physician has documented that the patient has HIV based on prior ELISA and western blot, or other approved diagnostic tests

PATIENT CHARACTERISTICS:

* Participants must be willing and able to sign an IRB-approved informed consent document

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected males and females age 18 and older with one of the three malignancy types studied with available diagnostic biopsy material
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ratner, MD, PhD, Principal Investigator — Washington University Siteman Cancer Center
Locations (14):
- United States (14):
  - Moores UCSD Cancer Center, La Jolla, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - John H. Stroger Hospital of Cook County, Chicago, Illinois
  - Louisiana State University Public Hospital, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pennsylvania - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Harborview Madison Clinic, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Results will be submitted to dBGaP

REFERENCES:
- See also: Clinicaltrials.gov summary of trial — https://clinicaltrials.gov/ct2/show/study/NCT01567722?term=AMC-083&rank=1

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical Cancer: Tissue collection for genomic sequencing from persons with a diagnosis of HIV and cervical cancer.
Period: Overall Study
Arm/Group | HIV-positive Diffuse Large B-cell Lymphoma Cases | HIV-positive Lung Cancer Cases | Cervical Cancer
Started | 93 | 19 | 2
Completed | 87 | 19 | 2
Not Completed | 6 | 0 | 0
Not completed — Not being able to get tissue for Central Pathology Review prior to the protocol closure date | 1 | 0 | 0
Not completed — Insufficient tissue available to satisfy the protocol requirements | 2 | 0 | 0
Not completed — Protocol closure by the OCG | 2 | 0 | 0
Not completed — Not enough tissue left for the tissue scrolls | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: HIV-positive persons age 18 and older with a diagnosis of a malignancy limited to the following diagnoses: any variant of diffuse large B cell lymphoma (DLBCL) except Burkitt's lymphoma, non-small cell lung malignancy or cervical cancer.
Groups:
- HIV Positive Cervical Cancer Cases: Tissue collection for genomic sequencing from persons with a diagnosis of HIV and cervical cancer.
- Total: Total of all reporting groups
Arm/Group | HIV-positive Diffuse Large B-cell Lymphoma Cases | HIV-positive Lung Cancer Cases | HIV Positive Cervical Cancer Cases | Total
Number analyzed (Participants) | 93 | 19 | 2 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.10 (10.86) | 61.42 (6.22) | 49.50 (7.78) | 51.97 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 2 | 21
  Male | 82 | 11 | 0 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 3 | 0 | 30
  Not Hispanic or Latino | 60 | 16 | 2 | 78
  Unknown or Not Reported | 6 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 32 | 10 | 2 | 44
  White | 51 | 6 | 0 | 57
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 3 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Collection of Tissue Specimen From Study Participants
Description: Summary of the specimens available by study arm
Time Frame: Study entry (prior to chemotherapy initiation)
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-positive Diffuse Large B-cell Lymphoma Cases | HIV-positive Lung Cancer Cases | HIV Positive Cervical Cancer Cases
Number analyzed (Participants) | 93 | 19 | 2
Participants
  Central pathology review | 85 | 18 | 2
  Formalin-fixed, paraffin-embedded tissue block for cental pathology review | 39 | 7 | 0
  Unstained slide from tissue | 65 | 12 | 2
  Specimen for Genomic sequence analysis | 71 | 16 | 2
  Snap frozen biopsy | 4 | 1 | 0
  Hematoxylin and eosin stained slide | 8 | 3 | 1
  Peripheral Blood Mononuclear Cells | 68 | 14 | 1
  Tissue core | 3 | 3 | 0
  Tissue scroll | 9 | 3 | 1
  Formalin-fixed, paraffin-embedded for genomic sequence analysis | 13 | 5 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data was not collected for this study..
Description: As a laboratory study involving only sample collection through routine clinical care and data abstraction, no adverse events was collected for this study.
Arm/Group | HIV-positive Diffuse Large B-cell Lymphoma Cases | HIV-positive Lung Cancer Cases | HIV Positive Cervical Cancer Cases
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT01567722/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT01567722/ICF_001.pdf